CLINICAL TRIAL: NCT07197125
Title: Prevalence of Anxiety and Depression Among Medical Students and Interns in Assiut University: Identifying Risk Factors and Academic Correlations
Brief Title: Psychological Burden of Anxiety and Depression Among Future Physicians: A Cross-sectional Study at Assiut University Faculty of Medicine
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Ali Khalaf Ahmed, resident at the Neuropsychiatry department, Assiut University
Other Study IDs: Anxiety and Depression
Record Dates: First submitted 2025-09-20; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Anxiety; Depression
Keywords: anxiety; depression
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The study population consists of undergraduate medical students and medical interns at Assiut Univer: Participants include medical students from first through fifth academic years at the Faculty of Medicine, Assiut University, along with first- and second-year interns (house officers) at Assiut University Hospital. This group represents a wide spectrum of the medical education process, from initial stages of training to early clinical practice.

SUMMARY:
A cross-sectional study will be conducted to assess the prevalence of anxiety and depression among medical students and interns at Assiut University, examining associated risk factors and their correlation with academic performance.

DETAILED DESCRIPTION:
This research aims to explore the prevalence of anxiety and depression among medical students and interns at Assiut University through a structured, anonymous Arabic self-administered questionnaire. The survey includes socio-demographic information, academic achievement, as well as standardized psychological assessment tools such as the Beck Depression Inventory (BDI) and Beck Anxiety Inventory (BAI). Data will be analyzed to determine overall prevalence rates, risk factors, and the trend of psychological morbidity across different academic grades and internship years. Special focus will be on identifying whether symptoms resolve, remain stable, or worsen during later academic years and internship. The study will provide essential insights into the mental health challenges faced by medical students and guide potential policies and student support interventions.

ELIGIBILITY:
Inclusion Criteria:

* Medical students at Assiut University (1st - 5th year)

Medical interns (1st and 2nd year) at Assiut University Hospital

Exclusion Criteria:

* Individuals with a previously diagnosed neurological disorder

Individuals with a previously diagnosed psychiatric disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants include medical students from first through fifth academic years at the Faculty of Medicine, Assiut University, along with first- and second-year interns (house officers) at Assiut University Hospital. This group represents a wide spectrum of the medical education process, from initial stages of training to early clinical practice. These students and interns are known to experience significant stress due to academic demands, examinations, and the transition to professional responsibilities, making them a particularly vulnerable group for psychological disorders.
Sampling Method: Probability Sample
Enrollment: 289 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of anxiety among medical students at Assiut University | baseline
  Measured using standardized Beck Anxiety Inventory (BAI) scales to determine the proportion of students experiencing symptoms of anxiety.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdel Wahed WY, Hassan SK. Prevalence and associated factors of stress, anxiety and depression among medical Fayoum University students. Alexandria J Med. 2017;53:77-84. doi:10.1016/j.ajme.2016.01.005